CLINICAL TRIAL: NCT03205423
Title: Medication Development for Opioid and Alcohol Abuse: Laboratory Study in Humans.
Brief Title: Medication Development for Opioid and Alcohol Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Sandra D. Comer, Professor of Neurobiology, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7476
Record Dates: First submitted 2017-03-08; First posted 2017-07-02 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two treatment conditions: gabapentin 0 mg or gabapentin 1800 mg/day first. Participants crossover to the 2nd gabapentin condition following a washout period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin 0 mg (Placebo Comparator): once daily at 8am
  Interventions: Drug: Gabapentin
- Gabapentin 1800 mg (Active Comparator): once daily at 8am
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Maintenance medication under investigation for its ability to alter the subjective and reinforcing effects of experimenter-administered doses of oxycodone and alcohol.

SUMMARY:
The present proposal will evaluate the ability of gabapentin maintenance to reduce the abuse liability of alcohol, oxycodone, and alcohol in combination with oxycodone in participants with both Opioid Use Disorder and Alcohol Use Disorder.

DETAILED DESCRIPTION:
Currently, the abuse of prescription opioid medications is a pervasive problem in the U.S. In addition, co-abuse of opioids and alcohol represents a significant problem from the perspective of increased toxicity and decreased success in treatment. Surprisingly few studies have examined the effects of combined administration of opioids and alcohol in humans, and no clinical studies have examined the reinforcing effects of this combination. The current 8-9-week inpatient study will systematically evaluate gabapentin because it shows promise for treating both opioid and alcohol use disorders (OUD and AUD). The guiding principle is that a medication's effects on positive subjective responses and reinforcing effects are the best laboratory procedures to date in predicting its clinical efficacy. We will examine the ability of gabapentin (0 mg or 1800 mg) to alter opioid-, alcohol-,and combined opioid/alcohol-mediated responses. Participants will meet DSM-5 criteria for moderate-severe OUD and be physically dependent on opioids. In addition, participants will meet DSM-5 criteria for moderate-severe AUD, but they will not be physically dependent on alcohol. All of the participants will be maintained on oral morphine throughout the study and different doses of gabapentin will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 criteria for moderate-severe opioid use disorder with physical dependence.
2. DSM-5 criteria for moderate-severe alcohol use disorder without physical dependence.
3. No current major mood, psychotic, or anxiety disorder.
4. Physically healthy.
5. Able to perform study procedures.
6. 21-59 years of age.
7. Normal body weight/Within 20% of body weight (for appropriate frame) according to 1983 Metropolitan Weight tables.
8. Current or history of illicit opioid use.
9. Current use of opioids in amounts and/or frequencies that meet or exceed those used in the proposed study (e.g., 3-4 tablets of a Rx opioid medication per day or 1-2 bags of heroin per day). Not seeking treatment for opioid use disorder (neutral attitude or not wanting treatment only).
10. Participants will consume alcohol at least 3 times per week (15 drinks per week for men and 8 drinks per week for women). In addition, they will drink alcohol and use opioids simultaneously.

Exclusion Criteria:

1. DSM-5 criteria for substance use disorder (moderate to severe) on drugs other than opioids, alcohol, nicotine or caffeine (must be less than 500 mg caffeine daily).
2. Participants requesting treatment.
3. Pregnancy or lactation.
4. Current or recent history of significant violent or suicidal behavior and/or suicidal/homicidal risk.
5. Cannot read or understand the self-report assessment forms unaided, or are so severely disabled that they cannot comply with the requirements of the study.
6. Elevated liver function tests (i.e., AST and ALT > 3 times the upper limit of normal) or impaired renal function (creatinine must be within normal limits).
7. Physical disorders that might make participation hazardous such as AIDS, cancer, hypertension (blood pressure > 140/90), uncontrolled diabetes, pulmonary hypertension or heart disease (please note that participants will be asked about previous visits to a cardiologist, chest pain, or strong palpitations; if these exist, they will be referred to a cardiologist and excluded unless cleared for participation by a cardiologist).
8. Current major Axis I psychopathology, other than OUD and AUD (e.g., mood disorder with functional impairment, schizophrenia), that might interfere with ability to participate in the study.
9. Sensitivity, allergy, or contraindication to opioids, alcohol, gabapentin or similar medications.
10. Taken an investigational drug within the past 30 days.
11. Current or history of chronic pain within the past 3 months.
12. Taking prescription psychotropic medications that would potentially interfere with study procedures.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D. Comer, PhD., Principal Investigator — New York State Psychiatric Institute / Columbia University Medical Center
Locations (1):
- New York State Psychiatric Institute in the Division on Substance Use Disorders, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castillo F, Harris HM, Lerman D, Bisaga A, Nunes EV, Zhang Z, Wall M, Comer SD. Clinical Implications of the Relationship Between Naltrexone Plasma Levels and the Subjective Effects of Heroin in Humans. J Addict Med. 2024 Mar-Apr 01;18(2):110-114. doi: 10.1097/ADM.0000000000001247. Epub 2023 Dec 20. PMID 38126709

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin (Active First): Gabapentin maintenance once daily at 8am for 8 weeks (1800 mg [(4 weeks) followed by 0 mg(4 weeks)]. In this trial, gabapentin is investigated for its ability to alter the subjective and reinforcing effects of experimenter-administered doses of oxycodone and alcohol.
- Gabapentin (Placebo First): Gabapentin maintenance once daily at 8am for 8 weeks (0 mg [(4 weeks) followed by 1800 mg (4 weeks)]. In this trial, gabapentin is investigated for its ability to alter the subjective and reinforcing effects of experimenter-administered doses of oxycodone and alcohol.
Period: Overall Study
Arm/Group | Gabapentin (Active First) | Gabapentin (Placebo First)
Started | 8 | 9
Completed | 7 | 6
Not Completed | 1 | 3
Not completed — Personal | 1 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Gabapentin (Within-Subjects): Participants are randomized to receive gabapentin once daily at 8am.
Arm/Group | Gabapentin (Within-Subjects)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 5
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Peak Positive Subjective Responses to Placebo.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: Assessed every 15 minutes following drug administration,for a total of 360 minutes. "Peak" drug effect is the highest rating throughout the entire testing session.
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 3.3 (.8) | 2.3 (.6)

2. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (30mg) + Low Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: Assessed every 15 minutes following drug administration, for a total of 360 minutes. "Peak" drug effect is the highest rating throughout the entire testing session.
Population: Participants who completed both the active and placebo phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 3.0 (.6) | 9.1 (1.2)

3. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (30mg) + High Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 6.7 (1.1) | 10.9 (1.3)

4. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (15mg) + High Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 6.3 (.9) | 9.7 (1.3)

5. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (15mg) + Low Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Gabapentin 1800: once daily at 8am
  Gabapentin: Maintenance medication under investigation for its ability to alter the subjective and reinforcing effects of experimenter-administered doses of oxycodone and alcohol.
Arm/Group | Gabapentin 0 mg | Gabapentin 1800
Number analyzed (Participants) | 13 | 13
units on a scale | 3.7 (.6) | 8.0 (1.1)

6. Primary Outcome: Peak Positive Subjective Responses to Low Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 4.1 (.7) | 11.4 (1.5)

7. Primary Outcome: Peak Positive Subjective Responses to High Alcohol Dose.
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 4.8 (.9) | 8.6 (1.2)

8. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (30mg)
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 2.7 (.7) | 5.3 (.9)

9. Primary Outcome: Peak Positive Subjective Responses to Oxycodone (15mg)
Description: Self-reported "High" measured on a 0-100 self-report visual analog scale. 0= Not-At-All 100=Extremely
Time Frame: as for outcome 2
Population: Participants who completed both the active and placebo gabapentin maintenance phases of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin 0 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 13 | 13
units on a scale | 1.9 (.4) | 4.7 (.9)

ADVERSE EVENTS:
Time Frame: Throughout the 4-week inpatient period
Groups:
- Gabapentin (0 mg, i.e., Placebo): Gabapentin maintenance (0 mg, i.e., placebo) once daily at 8 am for 4 weeks.
- Gabapentin (1800 mg i.e., Active): Gabapentin maintenance (1800 mg i.e., Active) once daily at 8 am for 4 weeks.
Arm/Group | Gabapentin (0 mg, i.e., Placebo) | Gabapentin (1800 mg i.e., Active)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (0 mg, i.e., Placebo) (N=17) | Gabapentin (1800 mg i.e., Active) (N=17)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03205423/Prot_SAP_ICF_002.pdf